CLINICAL TRIAL: NCT05311514
Title: Allogeneic Platelet Lysate Eye Drops for the Treatment of Severe Keratoconjunctivitis Sicca Resistant to Traditional Therapy in Patients With Chronic Ocular Graft-versus-host After Allogeneic Hematopoietic Stem Cell Transplantation.
Brief Title: Allogeneic Platelet Lysate Eye Drops for the Treatment of Severe Chronic Ocular Graft-versus-host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/21-n
Record Dates: First submitted 2021-10-01; First posted 2022-04-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Ocular Graft-versus-host Disease
Keywords: Chronic Graft-versus-host Disease; Ocular; Dry eye; Allogeneic stem cell transplantation; Platelet lysate; Eye drops
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic Platelet Lysate eye drops 50% (Experimental): Patients with ocular chronic severe graft versus host disease receive 50% allogeneic Platelet Lysate in the form of eye drops 6-8 times a day
  Interventions: Biological: Allogeneic platelet lysate eye drops
- Allogeneic Platelet Lysate eye drops 20% (Active Comparator): Patients with ocular chronic severe graft versus host disease receive 20% allogeneic Platelet Lysate in the form of eye drops 6-8 times a day
  Interventions: Biological: Allogeneic platelet lysate eye drops

INTERVENTIONS:
Biological: Allogeneic platelet lysate eye drops — Eye drops

SUMMARY:
The study evaluates the efficacy and safety of allogeneic platelet lysate eye drops in patients with severe ocular graft versus host disease refractory to conventional systemic and local treatments. The corneal staining, conjunctival hyperemia, tear film break up time,Schirmer test and ocular surface disease index will be evaluated before and after allogeneic platelet lysate treatment. The safety of allogeneic platelet lysate treatment will be also assessed.

DETAILED DESCRIPTION:
The corneal staining with fluorescein will be assessed using Oxford grading scale.

Tear film break up time is the time in seconds taken to appear first dry sport after complete blinking. Fluorescein is instilled into the patient tear film, the tear film is observed under cobalt blue illumination.Schirmer test will be performed without anesthesia. Conjunctival hyperemia will be graded from 0 to 2. The OSDI questinnaire will assess the impact of treatment on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Severe ocular chronic graft-versus-host disease (keratoconjunctivitis sicca) after allo-HSCT
* Schirmer test < 5mm\5min
* Tear Film Break-up Time < 5sec
* Corneal staining > II Gr (Oxford grading scale)
* Ocular Surface Disease Index (OSDI) >30
* Resistance to conventional therapy

Exclusion Criteria:

* Karnofsky <30%
* Other concomitant conditions, which does not allow to adequately assess the condition of the eye surface;
* Acute bacterial, viral or fungal infection of the eyes at the time of screening;
* Somatic or mental pathology that does not allow you to sign an informed consent;
* Keratoconjunctivitis sicca associated with an anomaly of the eyelids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Response of ocular chronic GVHD | 2 years
  Measured by 2015 NIH response criteria

SECONDARY OUTCOMES:
Ocular adverse events | 2 years
  Local ocular adverse events measured by CTCAE v5.0.
Tear film breakup time | 2 years
  Measured by fluorescein staining of the tear film
Area of epithelial damage | 2 years
  Measured by fluorescein staining of the ocular surface by the Oxford grading scale (grades 0-5 with increasing severity with higher grades)
Patient reported outcomes: severity of dry eye syndrome in patients with chronic ocular graft-versus-host and its impact on the quality of life based on 12 questions, score from 0 to 4. | 2 years
  Ocular Surface Disease Index (OSDI) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available upon request to the Pavlov Ethical Committee with the description of purposes and study plan according to local standard operating procedures.
Supporting Information: CSR
Time Frame: 15 years
Access Criteria: The individual participant data will be available upon request to the Pavlov Ethical Committee with the description of purposes and study plan according to local standard operating procedures.
URL: https://www.1spbgmu.ru/ru/92-glavnaya/nauka/sovety-i-komissii/eticheskij-komitet